CLINICAL TRIAL: NCT02655172
Title: Study on the Links Between Action and Perception in Schizophrenia, " Have a Good Grasp of the World "
Brief Title: Have a Good Grasp of the Worldthe World
Acronym: GRASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1508205; 2015-A01939-40 (Other: ANSM)
Record Dates: First submitted 2016-01-12; First posted 2016-01-13 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenic Disorders
Keywords: Schizophrenia, affordance,; perception-action binding,; stimulus-response-compatibility
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): patients suffering schizophrenic disorders and who will perform cognitive tasks + PANSS+ IQ
  Interventions: Other: cognitive tasks + PANSS+ IQ
- Control group (Active Comparator): healthy patients who will perform cognitive tasks
  Interventions: Other: cognitive tasks

INTERVENTIONS:
Other: cognitive tasks + PANSS+ IQ — Patients will perform different tasks: reaction time (Alert TEA, Zimmermann and Fimm, 2005), Edinburgh laterality questionnaire (Oldfield,1971), IQ test (IQ: PM38, Raven, 1960), and the PANSS (Positive and Negative Syndrome Scale (Kay et al., 1987) + the experimental task (affordance task with graspable device)
  Arms: Patients
Other: cognitive tasks — Healthy volunteers will perform only Edinburgh laterality questionnaire (Oldfield, 1971) + the experimental task (affordance task with graspable device).
  Arms: Control group

SUMMARY:
Brief Summary: In schizophrenia, dislocation of psychic functions involving a loss of contact with reality is frequently found. A fragmentation of motor and sensory perceptions could be held responsible. However, automatic integration between perception and action is the necessary condition to be in "relationship with the world." Affordance is the experimental link between object perception and potentially associated actions (Gibson, 1977, 1979) explored by Stimulus Response Compatibility (SRC) paradigm. With Tucker & Ellis sensory motor compatibility task (1998), with a modified response device (responses given with grasp), we study the impact of motor activation on these affordance effects. In this study, a group of controls will also be included in order to understand, as precisely as possible, the mechanisms involved (i.e., interference between the perception of the object and the response gesture).

DETAILED DESCRIPTION:
Schizophrenic patients will perform: Alert TEA, (Zimmermann and Fimm, 2005), Edinburgh laterality questionnaire (Oldfield, 1971), IQ test (IQ: PM38, Raven, 1960), and the PANSS (Positive and Negative Syndrome Scale, Kay et al., 1987). Controls will only perform the laterality questionnaire. Then all will perform the affordance task, in which photographs of 20 objects of everyday life, typically graspable with one hand, are presented in 4 orientations. Participants have to respond in a graspable device, as quickly as possible, if the object is presented upright or inverted.

ELIGIBILITY:
Inclusion Criteria:

* For patients:

  * a DSM-IV diagnosis of schizophrenia (men or women),
  * no change in antipsychotic medication and clinical status within four weeks prior to the study
* For patients and control group • Age ≥ 18 years et ≤ 55 years

Exclusion Criteria:

* History of head trauma,
* neurological disease with cerebral repercussion or not stabilized serious physical illness;
* psychotropic medication
* disorders related to the use of a psychoactive substance (abuse, dependence or withdrawal);

Exclusion Criteria:

* For patients:

  • IQ < 70
* For patients and control group

  * History of head trauma,
  * neurological disease with cerebral repercussion or not stabilized serious physical illness;
  * psychotropic medication
  * disorders related to the use of a psychoactive substance (abuse, dependence or withdrawal);

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
response time | day 1
  The gain provided by the compatible vs incompatible conditions (ms response time)

CONTACTS AND LOCATIONS:
Overall Officials: Anne GROSSELIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No